CLINICAL TRIAL: NCT05409300
Title: Phase II Trial Evaluating the Immunogenicity and Safety of BBIBP-CorV Vaccine in Adults in Guinea
Brief Title: Evaluation of the Immunogenicity and Safety BBIBP-CorV Vaccine for COVID-19 in Adults in Guinea
Acronym: CovicompareG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: CEPI (Other); Alliance for International Medical Action (Other); Centre National de Formation et de Recherche en Sante Rurale (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); APHP (Other); Agence Nationale de Sécurité Sanitaire de la Guinée (ANSS Guinée) (Unknown); Innovative clinical research network in vaccinology (IREIVAC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS0144S
Record Dates: First submitted 2022-03-28; First posted 2022-06-08 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Vaccine Adverse Reaction; Sars-CoV-2 Infection; Healthy Volunteer
Keywords: BBIBP-CorV; Elderly; SARS CoV 2 infected participants; Safety and immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — BIBP COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BBIBP-CorV (Experimental): Intramuscular administration of two doses of vaccine at 28 days (+/- 2 days) interval (0.5 mL/dose)
  Interventions: Biological: BBIBP-CorV

INTERVENTIONS:
Biological: BBIBP-CorV — Inactivated COVID19 vaccine, adjuvanted with aluminum hydroxide
  Other Names: Sinopharm

SUMMARY:
Phase II, non-randomized, open-label, comparative, single center national trial in Guinea, aimed to assess the humoral vaccine immune response induced by BBIBP-CorV vaccine in 200 adults aged between 18 and 45 years or 55 or older, one month after receiving the complete COVID-19 vaccination schedule.

DETAILED DESCRIPTION:
The main objective of this phase II trial is to evaluate the humoral immune response induced by the BBIBP-CorV vaccine in adults one month after complete vaccination regimen against SARS-CoV-2, comparing younger (up to 45 years old) and elderly (55+ years old) populations.

200 participants will be included. The age categories are 18 - 45 years, 55 - 64 years and 65+ years. The number of participants per age group will be distributed as follows 1:1:0,5. There will be no comparison between population on different vaccines.

Participants will receive two doses of BBIBP-CorV at 28 days interval. Vaccines will be administered intramuscular (0.5mL per injection)

Humoral vaccine immune responses, induced by BBIBP-CorV will be measured by ELISA at D0, M1, M2, M6, M12 and M24.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years old or 55 years and older
* Be eligible to receive one of the study vaccines as part of the trial
* Understand and agree to comply with study procedures (visits, telephone calls)
* Agree not to participate in any other vaccine study during the time of the study
* Give written informed consent prior to any examination performed as part of the trial

Exclusion Criteria:

* Age between 46 and 54 years old
* Positive SARS-CoV-2 antigenic test
* Positive SARS-CoV-2 PCR results less than 48 hours old
* History of infection by COVID-19 confirmed within 3 months prior to inclusion
* Symptoms compatible with COVID-19: sick or febrile participants (body temperature ≥ 38.0°C)
* Pregnant or breastfeeding woman
* Known chronic disease impacting the participant's immune response (uncured cancer, human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection)
* Anti-coagulant treatment
* Immunosuppressive treatment
* Contraindication to the proposed vaccine (according to RCP)
* Patient having received immunoglobulin or another blood product within 3 months prior to inclusion
* Previously received at least one injection of a SARS-CoV-2 vaccine
* A history of serious adverse vaccine reactions (anaphylaxis and associated symptoms such as rash, breathing difficulties, laryngeal edema, or a history of allergic reaction that may be exacerbated by a component of the SARS-CoV-2 vaccine)
* Any condition that, in the opinion of the investigator, may adversely affect the well-being of the participant and interfere with the purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 Spike IgG level | 1 month after complete vaccination schema
  Anti-SARS-CoV-2 Spike immunoglobulin G (IgG) level is measured using ELISA test

SECONDARY OUTCOMES:
Anti-SARS-CoV-2 specific IgG level | Day 0, Month 1, Month 2, Month 6, Month 12, and Month 24
  Anti-SARS-CoV-2 specific IgG level is measured using ELISA test
Anti-SARS-CoV-2 IgA and level | Day 0, Month 1, Month 2, Month 6, Month 12, and Month 24
  Anti-SARS-CoV-2 immunoglobulin A (IgA) level is measured using ELISA test
Anti-SARS-CoV-2 IgM level | Day 0, Month 1, Month 2, Month 6, Month 12, and Month 24
  Anti-SARS-CoV-2 immunoglobulin M (IgM) level is measured using ELISA test
Neutralizing antibody level for SARS-CoV-2 | Day 0, Month 1, Month 2, Month 6, Month 12, and Month 24
  Neutralizing antibody levels specific for SARS-CoV-2 and its variants (conventional in vitro neutralization and pseudo-neutralization assays)
Fluorospot tests (TH1, TH2, TH17, Cytotoxicity) | Day 0, Month 2, Month 6
  Fluorospot tests (Type 1,2,17 helper T cell (TH1, TH2, TH17), Cytotoxicity) Phenotyping of antigen-specific T cells by mass cytometry at Day 0 and Month 6 selected from the results of the Fluorospot test.
Mucosal SARS-CoV-2 specific antibody levels | Day 0, Month 1, Month 2, Month 6, Month 12
  Mucosal SARS-CoV-2 specific antibody levels by measuring IgA, IgM and IgG in saliva using specific ELISAs
Epitope profile | Day 0, Month 2
  Determination of epitope profile
B cell response to vaccine | Day 0, Month 2, Month 6
  Determination of repertoire of B cells (stereotype clonotype)
Measurement of ultrasensitive IgA and mucosal IgA and IgM functionality | Day 0, Month 1, Month 2, Month 6, Month 12, and Month 24
  Measurement of ultrasensitive IgA in saliva by Photoring assay Measurement of mucosal IgA and IgM functionality by SARS-CoV-2 mucosal IgA- and IgM-specific antibody-dependent cell-mediated cytotoxicity (ADCC) test
Rate of adverse events | Month 1 until Month 24
  Rate of adverse events of any grade attributable to the vaccine or vaccination occurring between Month 1 and Month 24
SARS-CoV-2 infection | Day 0 until Month 24
  Occurrence of confirmed COVID-19 cases during participant follow-up

OTHER OUTCOMES:
Measurement of specific B memory cells | Day 0, Month 2, Month 6, Month 12
  Measurement of specific B memory cells (Elispot B)
Measurement of specific T cell response | Day 0, Month 12
  Measurement of specific T cell response (Cytof analysis)
Identification of predictive determinants of vaccine response | Month 24
  Identification of pre-existing immunity against other coronaviruses or respiratory pathogens, immunosenescence profile, transcriptomic, metabolomic and proteomic analysis, cytokine profile (IFNa), immune cell phenotype
Quantitative measures | Day 0 until Month 24
  Quantitative measures: Number of participants recruited, number of follow-up visits carried out, proportion of participants satisfied with the vaccine received

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, Study Chair — Innovative clinical research network in vaccinology (I-REIVAC); Abdoul Habib Beavogui, Principal Investigator — Centre National de Formation et de Recherche en Santé Rurale (CNFRSR)
Locations (2):
- Guinea (2):
  - Centre de recherche de Landreah, Conakry
  - Palais du Peuple, Conakry

IPD SHARING:
Plan to Share IPD: Yes